CLINICAL TRIAL: NCT04870034
Title: Perioperative Analysis of Binimetinib and Palbociclib in RAS-Driven Tumors
Brief Title: Binimetinib and Palbociclib Before Surgery for the Treatment of Operable KRAS-Positive Lung, Colorectal, or Pancreatic Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Issues recruiting
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 797920; NCI-2021-02908 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 797920 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Carcinoma; Lung Adenocarcinoma; Malignant Solid Neoplasm; Pancreatic Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma of Lung; Pancreatic Neoplasms | interventions — binimetinib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (palbociclib, binimetinib) (Experimental): Patients receive palbociclib PO QD and binimetinib PO BID for 14 days in the absence of disease progression or unacceptable toxicity. Within 1 week after last dose of study medication, patients undergo surgery.
  Interventions: Drug: Binimetinib; Drug: Palbociclib; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This early phase I trial studies the direct effects on cancer cells of the drugs binimetinib and palbociclib, in patients with KRAS-positive lung, colorectal, or pancreatic cancer that can be removed by surgery (operable). Binimetinib and palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving binimetinib and palbociclib may halt the growth of cancer cells and improve access of the immune system cells, a patient's own cells that fight infection and cancer, into the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the on-target efficacy of binimetinib and palbociclib in patients with operable RAS-mutant lung adenocarcinoma, colorectal, or pancreatic cancer.

SECONDARY OBJECTIVES:

I. Correlative analysis of gene expression analysis. II. Define immune subsets within the pre and post-treatment tumor tissue.

OUTLINE:

Patients receive palbociclib orally (PO) once daily (QD) and binimetinib PO twice daily (BID) for 14 days in the absence of disease progression or unacceptable toxicity. Within 1 week after last dose of study medication, patients undergo surgery.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients with verified and operable KRAS-positive mutant lung adenocarcinoma, colorectal, or pancreatic cancer
* Have available diagnostic, pre-treatment archival tumor tissue
* Medically fit for surgical resection
* Absolute neutrophil count (ANC) >= 1500/ uL
* Hemoglobin (Hgb) >= 9 g/dL
* Platelet count >= 100,000/uL
* Total bilirubin =< 1.5 x ULN (upper limit of normal)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x ULN
* Creatinine clearance > 60 mL/min (Cockcroft-Gault Equation)
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Ability to swallow and retain oral medication
* Female participants of childbearing potential must agree to use methods of contraception that are highly effective or acceptable, and to not donate ova from screening until 30 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male participants must agree to use methods of contraception that are highly effective or acceptable, and to not donate sperm from screening until 90 days after the last dose of study drug
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior therapy with a CDK4/6 (e.g. palbociclib, ribociclib) or MEK inhibitor (e.g., binimetinib, trametinib, cobimetinib)
* Participants who have had any other systemic anticancer therapy within 2 weeks prior to entering the study
* Is currently participating in a study and receiving an investigational agent; has received an investigational agent within 14 days prior to start of study treatment
* Participants who have undergone major surgery =< 6 weeks prior to start of study treatment or who have not recovered from side effects of such procedure
* Patient has not recovered to =< grade 1 from toxic effects of prior therapy before starting study treatment. Note: Stable chronic conditions (=< grade 2) that are not expected to resolve (such as neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies) are exceptions and may enroll
* Uncontrolled or symptomatic brain metastases or leptomeningeal carcinomatosis that are not stable, require steroids, are potentially life-threatening or have required radiation within 28 days prior to starting study drug. Note: Patients with previously treated brain metastases may participate provided they are stable (e.g., without evidence of progression by radiographic imaging for at least 28 days before the first dose of study treatment and neurologic symptoms have returned to baseline), and have no evidence of new or enlarging brain metastases or central nervous system (CNS) edema, and does not require steroids at least 7 days before the first dose of study treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Impaired cardiovascular function or clinically significant cardiac diseases including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to screening
  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2)
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition scan (MUGA) or echocardiography (ECHO)
  * Uncontrolled hypertension defined as persistent systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia)
  * Baseline corrected QT (QTc) interval >= 480 ms
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of binimetinib or palbociclib (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (=< 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs
* Patients who have neuromuscular disorders that are associated with elevated creatine kinase (CPK) (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* Current use of a prohibited medication (including herbal medications, supplements, or foods) or use of a prohibited medication =< 1 week prior to the start of study treatment
* History of or cerebrovascular events =< 12 weeks prior to the first dose of study treatment
* History of pulmonary embolism (PE) with hemodynamic instability =< 12 weeks prior to first dose of study treatment. Note: Patients with PE that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of therapeutic anticoagulants for at least 4 weeks. Also, patients with deep vein thrombosis on stable dose of therapeutic anticoagulants for at least 4 weeks are allowed to participate in the study
* Concurrent or previous other malignancy that requires active anticancer therapy
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

  * Note: Patients with laboratory evidence of cleared HBV or HCV infection may be enrolled
  * Note: Patients with no prior history of HBV infection who have been vaccinated against HBV and who have a positive antibody against hepatitis B surface antigen as the only evidence of prior exposure may be enrolled
* Known history of acute or chronic pancreatitis =< 6 months prior to enrollment
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) =< 12 months prior to enrollment
* Known hypersensitivity to the components of study drugs or its analogs
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study
* The following special populations will not be included in the study:

  * Cognitively impaired adults/adults with impaired decision-making capacity
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Ki67 labeling index of > 70% | Up to 30 days post treatment
  Pathologic response by change in Ki-67% from pre and surgical biopsies
Incidence of adverse events | Up to 30 days post-treatment
  Toxicities and adverse events (as per Common Terminology Criteria for Adverse Events version 5.0) will be summarized by attribution and grade using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Gene expression analysis | Up to 30 days post-treatment
  Correlative analysis of gene expression analysis will focus on suppression of MEK and CDK4/6 regulated genes and induction of gene expression programs related to antigen presentation and inflammation.
Immune subsets within the pre and posttreatment tumor tissue | Up to 30 days post-treatment
  Multispectral imaging will be employed to define immune subsets within the pre and posttreatment tumor tissue with an emphasis on approaches to exploit the response to drug with immunologically active agents.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States